CLINICAL TRIAL: NCT02234219
Title: Comparison of Circular(Soave) and Heart-shaped Anastomosis in Hirschsprung's Disease: A Prospective Multicenter Randomized Controlled Trial
Brief Title: Comparison of Circular(Soave) and Heart-shaped Anastomosis in Hirschsprung's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jiexiong Feng, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anastomosis in Hirschsprung
Record Dates: First submitted 2014-08-27; First posted 2014-09-09 (Estimated); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart-shaped anastomosis (Experimental): Heart shaped anastomosis
  Interventions: Procedure: Heart-shape anastomosis
- Circle anastomosis (Active Comparator): Soave anastomosis
  Interventions: Procedure: Soave anastomosis

INTERVENTIONS:
Procedure: Heart-shape anastomosis — a new operation approach for Hirschsprung disease
  Arms: Heart-shaped anastomosis
Procedure: Soave anastomosis — traditional approach for Hirschsprung disease
  Arms: Circle anastomosis

SUMMARY:
Comparison of Circular(Soave)and Heart-shaped Anastomosis in Hirschsprung's disease.

DETAILED DESCRIPTION:
At present, the treatment for children with HSCR is still surgery. The basic treatment principles of all surgical procedures commonly used in the world include confirming the location of the transitional zone between the intestinal tube with and without ganglion cells, removing the intestinal segment without ganglion cells, and reconstructing the digestive tract by anastomosis of the intestinal segment with ganglion cells with the anus or rectum. Intact anal receptors and autonomic internal sphincter control are essential for autonomic bowel control, and the integrity of the internal sphincter directly affects the occurrence of soilage and fecal incontinence after surgery. Therefore, how to deal with the internal sphincter during the operation, so as to avoid the recurrence of constipation caused by the spasm of the internal sphincter after the operation, and to retain the function of the internal sphincter for defecation control has been the focus of research.

In the 1980s, Professor Wang Guo, based on the experience of previous researchers, innovated the "heart-shaped anastomosis", which is a surgical procedure in which the dorsal rectum is split longitudinally to the dentate line without removing the internal sphincter, and then the normal colon is drawn out to make an oblique anastomosis with the rectoanal canal. A retrospective single-center follow-up of nearly 100 cases of "heart-shaped anastomosis" over a period of 20 years found that compared with traditional end-to-end colorectal anastomosis, patients with "heart-shaped anastomosis" had a significantly lower rate of fecal fouling and a long-term Bowel function score (Bowel function score, bowel function score). BFS) and Quality of Life-BREF (QLB) were also significantly improved compared with the traditional operation (P<0.05), and no other adverse events occurred. This study aims to determine the optimal surgical procedure for HSCR by a prospective, multicenter controlled study comparing the "heart-shaped anastomosis" with the commonly used Soave procedure.

In summary, this project will compare the application of "heart-shaped anastomosis" and traditional surgery for children with HSCR before operation, and comprehensively evaluate the advantages of "heart-shaped anastomosis" for defecation control from morphology to electrophysiological function through postoperative follow-up, combined with anorectal manometry.

ELIGIBILITY:
Inclusion Criteria:

1. Age<14 years
2. Hirschsprung's disease diagnosed by biopsy
3. Surgical indication

Exclusion Criteria:

1. Age>14 years
2. Not Hirschsprung's disease
3. Surgical contraindication

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
bowel function score | 2 years
  Ability to control bowel movements, Feeling before bowel movement, Soiling, Defecation frequency, Constipation, Social problem

SECONDARY OUTCOMES:
rate of postoperative complication | 1month/6 month/12 month/2 years
  HAEC/anastomosis leakage/soiling/constipation recurrence et al.
rate of reoperation | 1month/6 month/12 month/2 years
  rate of reoperation
rate of readmission | 1month/6 month/12 month/2 years
  rate of readmission
bowel function score | 1 month/6 month/12 month
  Ability to control bowel movements, Feeling before bowel movement, Soiling, Defecation frequency, Constipation, Social problem

CONTACTS AND LOCATIONS:
Overall Officials: Jiexiong Feng, MD., Principal Investigator — Department of Pediatric surgery, Tongji hospital, HUST, Wuhan
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China